CLINICAL TRIAL: NCT00866086
Title: Study of Automated Abdominal Compression Device and Screw Based Abdominal Compression Devices During Stereotactic Body Radiation Therapy of Lung Tumors
Brief Title: Comfort Level of Two Abdominal Compression Methods Used to Hold Patients Still While Undergoing Stereotactic Body Radiation Therapy for Lung Tumors
Status: Terminated | Phase: Phase 1 | Type: Interventional
Why Stopped: low accrual
Sponsor: University of Texas Southwestern Medical Center (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: SCCC-122008-012; CDR0000634652 (Registry Identifier: PDQ (Physician Data Query))
Record Dates: First submitted 2009-03-19; First posted 2009-03-20 (Estimated); Last update posted 2020-08-20 (Actual); Status verified 2019-03

CONDITIONS: Lung Cancer
Keywords: stage I non-small cell lung cancer; stage II non-small cell lung cancer; stage IIIA non-small cell lung cancer; stage IIIB non-small cell lung cancer; stage IV non-small cell lung cancer; recurrent non-small cell lung cancer; pulmonary carcinoid tumor; extensive stage small cell lung cancer; limited stage small cell lung cancer; recurrent small cell lung cancer
MeSH Terms: conditions — Lung Neoplasms; Carcinoma, Non-Small-Cell Lung; Small Cell Lung Carcinoma

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

INTERVENTIONS:
Other: questionnaire administration
Procedure: computed tomography
Radiation: radiation therapy treatment planning/simulation

SUMMARY:
RATIONALE: Stereotactic body radiation therapy may be able to send x-rays directly to the tumor and cause less damage to normal tissue. Abdominal compression methods that hold the body and the tumor from moving during treatment may permit radiation therapy to kill more tumor cells. This study is looking at the comfort level of two abdominal compression methods in patients with lung tumors undergoing stereotactic body radiation therapy.

PURPOSE: This phase I trial is studying the comfort level of two abdominal compression methods used to hold patients still while undergoing stereotactic body radiation therapy for lung tumors.

DETAILED DESCRIPTION:
OBJECTIVES:

Primary

* To evaluate comfort associated with the existing screw-based abdominal compression device and the new automated abdominal compression device in patients with lung tumors undergoing stereotactic body radiotherapy.

Secondary

* To evaluate tumor motion in patients using these devices.

OUTLINE: This is a multicenter study.

Patients undergo fluoroscopic assessment of tumor motion with a screw-based abdominal compression device. Patients then undergo non-contrast 4D-CT imaging with the screw-based abdominal compression device followed by contrast 4D-CT imaging with an automated abdominal compression device.

Immediately after stereotactic body radiotherapy simulation, patients complete a questionnaire to assess the overall level of comfort of each abdominal-compression device.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* All lung patients from the University of Texas Southwestern Medical Center, Parkland Health and Hospital System, and Richardson Regional Cancer Center scheduled to receive stereotactic body radiotherapy simulation
* Must have initial pre-compression lung tumor motions with respiration > 1 cm

PATIENT CHARACTERISTICS:

* Negative pregnancy test

PRIOR CONCURRENT THERAPY:

* Concurrent participation in other protocols allowed

Ages: 18 Years to 120 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10 (Estimated)
Dates: Start 2009-02 (Actual); Primary Completion 2009-06 (Actual); Study Completion 2009-09 (Actual)

PRIMARY OUTCOMES:
Patient comfort score | 10 years

SECONDARY OUTCOMES:
Tumor motion as measured by screw-based and automated abdominal compression devices and 4D-CT imaging | 10 years

CONTACTS AND LOCATIONS:
Overall Officials: Robert D. Timmerman, MD, Principal Investigator — Simmons Cancer Center
Locations (1):
- Simmons Comprehensive Cancer Center at University of Texas Southwestern Medical Center - Dallas, Dallas, Texas, United States

IPD SHARING:
Plan to Share IPD: No